CLINICAL TRIAL: NCT03209869
Title: Treatment of Relapsed or Refractory Neuroblastoma and Osteosarcoma With Ex-Vivo Expanded and Activated Haploidentical NK Cells and Hu14.18-IL2
Brief Title: Treatment of Relapsed or Refractory Neuroblastoma and Osteosarcoma With Expanded Haploidentical NK Cells and Hu14.18-IL2
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: resources limited due to COVID-19
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Solving Kids' Cancer (Other); Midwest Athletes Against Childhood Cancer, Inc. (MACC Fund) (Unknown); Wade's Army (Unknown); The Catherine Elizabeth Blair Memorial Foundation / GWCF (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW16009; P30CA014520 (NIH); 2016-1195 (Other: Institutional Review Board); A536755 (Other: UW Madison); SMPH/PEDIATRICS/PEDIATRICS (Other: UW Madison); NCI-2017-01267 (Registry Identifier: NCI Trial ID); Protocol V12 01/30/2021 (Other: UW Madison)
Record Dates: First submitted 2017-06-13; First posted 2017-07-06 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Neuroblastoma; Relapsed Neuroblastoma; Recurrent Neuroblastoma; Osteosarcoma
MeSH Terms: conditions — Neuroblastoma; Osteosarcoma | interventions — lorukafusp alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): All subjects will receive Ex vivo Expanded and Activated Haploidentical Donor NK Cells + hu14.18-IL2
  Interventions: Biological: Ex vivo Expanded and Activated Haploidentical Donor NK Cells; Biological: Hu14.18-IL2

INTERVENTIONS:
Biological: Ex vivo Expanded and Activated Haploidentical Donor NK Cells — Haploidentical donor NK cells that are expanded and activated under current GMP conditions using K562-mbIL15-41BBL.
  Other Names: EANK cells
Biological: Hu14.18-IL2 — The immunocytokine, hu14.18-IL2, is a fusion protein comprised of one molecule of the anti-GD2 humanized monoclonal antibody, hu14.18, fused to two molecules of the cytokine, interleukin-2.
  Other Names: Immunocytokine

SUMMARY:
Subjects with relapsed or refractory neuroblastoma and osteosarcoma will receive ex-vivo expanded and activated natural killer (NK) cells from a haploidentical donor in conjunction with the immunocytokine, hu14.18-IL2.

DETAILED DESCRIPTION:
Natural Killer cells, a type of white blood cell, circulate around the body and kill abnormal cells (cells that are malignant, damaged or infected with virus). Sometimes cancer cells adapt to the body's own NK cells and are able to avoid being killed by them. This clinical trial uses two strategies to overcome the cancer cells' ability to avoid NK cell-mediated death.

The first strategy involves giving NK cells from another individual to the patient (in other words, donor- or haploidentical-NK cells). This is done because NK cells from an individual who is haploidentical (half-matched genetic make-up) are still able to effectively kill the cancer cells. Unfortunately, only a limited number of NK cells can be obtained from a donor. So, to increase the number of cancer-killing NK cells that will be given to the patient, the donor NK cells will first be grown in a sterile laboratory environment and allowed to multiply many-fold before they are infused into the patient. This growing process also activates the donor NK cells, which increases their ability to kill cancer cells.

The second strategy to overcome the cancer cells' ability to avoid NK cell-mediated death is to administer the immunocytokine, hu14.18-IL2, every day for seven days after infusion of the donor NK cells. The antibody portion (hu14.18) of the immunocytokine molecule "flags" the neuroblastoma cells for destruction by NK cells and the cytokine portion (IL2) further activates the NK cells (as well as other anti-tumor immune effector cells).

Since the donor NK cells are from a haploidentical individual, they are different enough to be recognized as foreign cells and will be killed immediately ("rejected") by the patients own immune system unless the immune system is restrained. So, to allow the donor NK cells time to kill neuroblastoma cells before they are "rejected", a chemotherapy regimen is first given to the patient to temporarily restrain the patient's own immune system. This also allows "room" for the donor NK cells to live, multiply and function.

Four courses of treatment are planned for each subject. Each course of treatment will be approximately one month long and involves a week of chemotherapy followed by infusion of donor NK cells. Beginning the day after the donor NK cell infusion, hu14.18-IL2 is infused over four hours for seven consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory neuroblastoma
* Relapsed or refractory Osteosarcoma
* Karnofsky/Lansky performance score > 50
* Life expectancy ≥ 4 months
* Creatinine clearance or radioisotope GFR ≥ 60 ml/min/1.73m2 OR serum creatinine within normal limits based on age and gender
* ANC ≥ 750/µL
* Platelet count ≥ 50,000/µL
* Hemoglobin ≥ 8 g/dL
* Total bilirubin ≤ 1.5 x upper limit of normal for age
* ALT (SCPT) ≤ 5 x upper limit of normal for age
* Shortening fraction of ≥ 27% by echocardiogram OR Ejection fraction of ≥55% by MUGA
* No evidence of dyspnea at rest
* Pulse oximetry > 94% on room air
* If PFTs performed, FEV1/FVC must be > 60%
* All Osteosarcoma patients must have PFTs performed
* CNS toxicity ≤ Grade 2
* Patients with seizure disorders may be enrolled if seizures are well controlled on anticonvulsant therapy
* > 100 days after autologous stem cell infusion following myeloablative therapy
* ≥ 2 weeks since chemotherapy
* ≥ 7 days since anti-neoplastic, non-myelosuppressive biologic agent (or extended for agents known to have adverse events beyond the 7- day period)
* ≥ 2 weeks for local palliative XRT
* ≥ 6 months if prior craniospinal axis XRT (> 50%)
* ≥ 6 months if > 50% radiation of pelvis
* ≥ 6 weeks after therapeutic 131I-MIBG
* ≥ 6 weeks since thoracotomy
* Informed consent obtained (patient or legal representative)
* Women of reproductive potential must have negative pregnancy test and be willing to use effective birth control method
* Suitable haploidentical donor must be available

Exclusion Criteria:

* Prior history of ventilator support related to lung injury, except for immediately following thoracotomy
* Symptomatic pleural effusions or ascites
* <6 weeks from thoracotomy and <2 weeks from other major surgery
* History of anaphylaxis while receiving prior anti-GD2 therapy
* Pregnant
* HIV infection
* Heart failure or uncontrolled cardiac rhythm disturbance
* Active infection
* Prior organ allograft
* Prior allogeneic bone marrow or peripheral blood stem cell transplant
* Significant serious intercurrent illnesses expected to interfere with the antitumor effect of treatment or to significantly increase the severity of toxicities experienced from treatment
* Any mental or physical condition, in the opinion of the PI (or PI designee), which could interfere with the ability of the subject (or the only parent or legal guardian available to care for the subject) to understand or adhere to the requirements of the study.
* Enrollment in any other treatment study from screening up to 28 days after the last treatment on this study (unless PI judges such enrollment would not interfere with endpoints of this study)

Ages: 7 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of treatment-emergent adverse events of treatment with AENK cells and hu14.18-IL2 | up to 28 days after final dose of EA-NK cells or hu14.18-IL2, whichever occurs last
  Safety will be assessed by quantifying adverse events ≥ grade 3, using CTCAE (v.5), with certain pre-defined exceptions based on known, transient, reversible, clinically manageable toxicities of the chemotherapy and hu14.18-IL2.
Safety: Incidence of any grade acute or chronic GVHD | up to 21 days after final dose of EA-NK cells or hu14.18-IL2, whichever occurs last
  Safety will be assessed by monitoring for any grade acute or chronic GVHD.

SECONDARY OUTCOMES:
Efficacy: Progression free survival | up to12 months after final dose of EA-NK cells or hu14.18-IL2, whichever occurs last
  The time elapsed from initial EANK cell infusion until disease progression or death or study censure 12 months after final dose of immunotherapy
Efficacy: Overall survival | up to12 months after final dose of EA-NK cells or hu14.18-IL2, whichever occurs last
  The time from initial EANK cell infusion until death from any cause or study censure 12 months after final dose of immunotherapy
Efficacy: Objective tumor response (SD + CR + PR) | up to12 months after final dose of EA-NK cells or hu14.18-IL2, whichever occurs last
  The anti-tumor effect of treatment will be assessed by quantifying the number of subjects who achieve stable disease, complete remission and partial remission
Longevity of EA-NK cells in vivo | 28 days
  Evaluating the survival of EA-NK cells in the subject using flow cytometric analysis of donor-only antigens
Immunocytokine (hu14.18-IL2) serum levels given as daily infusions for 7 consecutive days | up to 28 days after last hu14.18-IL2 infusion
  Hu14.18-IL2 serum levels will be assessed using ELISA
Immunogenicity of hu14.18-IL2 given as daily infusions for 7 consecutive days | up to 28 days after last hu14.18-IL2 infusion
  Measurement of anti-hu14.18-IL2 antibodies (HAHA) using ELISA
Proportion and absolute numbers of NK and T cell subsets | up to 22 days after the third EANK cell infusion for subjects in Cohort A and up to 22 days after the second EANK cell infusion for subjects in Cohort B
  NK and T cell subsets will be evaluated using flow cytometric assessment of cell phenotype expressed as percentages of larger cell subsets and absolute numbers.
EANK cell survival in vivo | up to 22 days after the third EANK cell infusion for subjects in Cohort A and up to 22 days after the second EANK cell infusion for subjects in Cohort B
  The longevity of EANK cells in vivo (i.e., after infusion) will be assessed by evaluating donor-specific HLA markers present on NK cells using flow cytometry
NK cell activity | up to 22 days after the third EANK cell infusion for subjects in Cohort A and up to 22 days after the second EANK cell infusion for subjects in Cohort B
  The functional status of NK cells will be measured: 1) indirectly by assessing NK activation receptor expression and NK exhaustion marker expression using flow cytometric analyses and 2) directly by measuring the ability of NK cells to kill tumor cells in vitro

CONTACTS AND LOCATIONS:
Overall Officials: Ken DeSantes, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center; UW Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UW Carbone Cancer Center Home Page — http://www.uwhealth.org/uw-carbone-cancer-center/cancer/10252